CLINICAL TRIAL: NCT00620256
Title: Comparison of Safety and Efficacy of Al-37807 Ophthalmic Suspension vs. Timolol Gel Forming Solution and Vehicle, All Dosed Concomitantly With Xalatan in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Adjunctive Study of AL-37807 Ophthalmic Suspension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-07-05
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AL-37807 (Experimental): AL-37807 ophthalmic suspension, 0.1%, one drop in the study eye(s) at 8 AM, with latanoprost ophthalmic solution, one drop in the study eye(s) at 8 PM, for four weeks
  Interventions: Drug: AL-37807 ophthalmic suspension, 0.1%; Drug: Latanoprost ophthalmic solution
- Timolol (Active Comparator): Timolol gel forming solution, 0.5%, one drop in the study eye(s) at 8 AM, with latanoprost ophthalmic solution, one drop in the study eye(s) at 8 PM, for four weeks
  Interventions: Drug: Timolol gel forming solution, 0.5%; Drug: Latanoprost ophthalmic solution
- AL-37807 vehicle (Placebo Comparator): AL-37807 ophthalmic solution vehicle, one drop in the study eye(s) at 8 AM, with latanoprost ophthalmic solution, one drop in the study eye(s) at 8 PM, for four weeks
  Interventions: Drug: AL-37807 ophthalmic suspension, 0.1%; Other: AL-37807 ophthalmic solution vehicle; Drug: Latanoprost ophthalmic solution

INTERVENTIONS:
Drug: AL-37807 ophthalmic suspension, 0.1%
  Arms: AL-37807; AL-37807 vehicle
Drug: Timolol gel forming solution, 0.5%
  Arms: Timolol
Other: AL-37807 ophthalmic solution vehicle
  Arms: AL-37807 vehicle
Drug: Latanoprost ophthalmic solution
  Other Names: XALATAN

SUMMARY:
The purpose of the study is to compare the safety and intraocular pressure-lowering efficacy of AL-37807 ophthalmic suspension vs. Timolol gel forming solution vs. AL-37807 vehicle, all dosed concomitantly with Xalatan, in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Open-angle glaucoma
* Ocular hypertension
* Must have been on Xalatan for at least 3 months
* VA not worse than 0.60
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Age related
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in intraocular pressure | Baseline, up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center at 1-888-451-3937, Fort Worth, Texas, United States